CLINICAL TRIAL: NCT01407276
Title: An Open-Label, Two-Part, Single-Dose Study to Investigate the Pharmacokinetics, Safety and Tolerability of MK-3102 in Patients With Impaired Renal Function
Brief Title: A Study of Omarigliptin (MK-3102) in Participants With Impaired Renal Function (MK-3102-009)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3102-009
Record Dates: First submitted 2011-07-29; First posted 2011-08-02 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Chronic Renal Insufficiency; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part 1: Mild Renal Impairment (Panel A) (Experimental)
  Interventions: Drug: Omarigliptin
- Part 1: Control to Match Panel A (Panel B) (Experimental)
  Interventions: Drug: Omarigliptin
- Part 1: Moderate Renal Impairment (Panel C) (Experimental)
  Interventions: Drug: Omarigliptin
- Part 1: Control to Match Panel C (Panel D) (Experimental)
  Interventions: Drug: Omarigliptin
- Part 1: Severe Renal Impairment (Panel E) (Experimental)
  Interventions: Drug: Omarigliptin
- Part 1: Control to Match Panel E (Panel F) (Experimental)
  Interventions: Drug: Omarigliptin
- Part 2: End-stage Renal Disease needing hemodialysis (Panel G) (Experimental)
  Interventions: Drug: Omarigliptin
- Part 2: Control to Match Panel G (Panel H) (Experimental)
  Interventions: Drug: Omarigliptin

INTERVENTIONS:
Drug: Omarigliptin — Single oral dose of 3 mg (3 x 1-mg capsules)
  Other Names: MK-3102

SUMMARY:
This is a 2-part study in participants with renal impairment and matched healthy participants to investigate the effect of impaired renal function on the plasma and urine levels of omarigliptin (MK-3102) after taking a single 3 mg dose by mouth.

DETAILED DESCRIPTION:
In Part I, three panels of 6 participants each will be enrolled with varying degrees of renal disease (mild, moderate, or severe renal impairment) based on their estimated glomerular filtration rate (eGFR). Each of these panels will be matched with a corresponding panel of equal number of healthy, age-, race-, BMI- and gender-matched control participants. All panels will receive a single oral dose of 3-mg omarigliptin, followed by plasma sampling and urine collection. In Part II, 6 participants with end stage renal disease (ESRD) requiring hemodialysis will receive a single 3-mg oral dose of omarigliptin immediately following hemodialysis (HD) (Period 1) and 2 hours prior to HD (Period 2).There will be approximately 1 month between Period 1 and Period 2. A corresponding panel of equal number, healthy matched control subjects (age, race, BMI, gender) will also receive a single 3 mg dose by mouth. Omarigliptin dose administration will be followed by plasma sampling for both panels.

ELIGIBILITY:
Inclusion Criteria:

Impaired Renal Function Subjects:

* Females of reproductive potential must have a negative pregnancy test and agree to use 2 methods of birth control
* Diagnosis of renal insufficiency based on estimated glomerular filtration rate (eGFR) calculated using the Modification of Diet in Renal Disease (MDRD) equation

Healthy Subjects:

* Females of reproductive potential must have a negative pregnancy test and agree to use 2 methods of birth control;
* In general good health

Exclusion Criteria:

Impaired Renal Function Subjects:

* Is mentally or legally incapacitated
* Has rapidly fluctuating renal function or has demonstrated or suspected renal artery stenosis
* History of significant endocrine (other than Type 2 diabetes), gastrointestinal, cardiovascular, hematological, immunological, respiratory, or genitourinary diseases
* History of stroke, chronic seizures or major neurological disease
* Uncontrolled Type 2 diabetes or history of Type 1 diabetes or ketoacidosis
* History of cancer (Some exceptions apply)
* Regular user of barbiturates or sleep aides
* Consumes excessive amounts of alcohol (more than 2 drinks/day)
* Consumes excessive amounts of caffeinated beverages (more than 6/day)
* Has had major surgery or has lost or donated 1 unit of blood within 4 weeks
* Has a history of significant multiple and/or severe allergies
* Current or history of illicit drug abuse
* Nursing mothers

Healthy Subjects:

* Is mentally or legally incapacitated;
* Has a history of stroke, chronic seizures, or major neurological disorder
* Renal impairment
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, immunological, respiratory, or genitourinary diseases
* Hypoglycemia, glucose intolerance, Type 1 or Type 2 diabetes, or ketoacidosis
* History of cancer (Some exceptions apply)
* Regular user of barbiturates or sleep aides
* Consumes excessive amounts of alcohol (more than 2 drinks/day)
* Consumes excessive amounts of caffeinated beverages (more than 6/day)
* Has had major surgery or has lost or donated 1 unit of blood within 4 weeks
* Has a history of significant multiple and/or severe allergies
* Current or history of illicit drug abuse
* Nursing mothers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-08-08 (Actual); Primary Completion 2012-03-23 (Actual); Study Completion 2012-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis Links — http://www.merck.com/clinical-trials/study.html?id=3102-009&kw=3102-009&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One healthy matched control participant withdrew consent for study participation on Day 15; this participant was replaced. Thus, a total of 49 participants were in the study.
Groups:
- Part 1: Mild Renal Impairment (Panel A): Participants with estimated glomerular filtration rate (eGFR) ≥60 - <80 mL/min/1.73 m² were enrolled in the Mild Renal Impairment group.
- Part 1: Control to Match Panel A (Panel B): Participants with eGFR >/= 80 mL/min/1.73 m² were matched by age, gender, race, and body mass index (BMI) to participants in Panel A.
- Part 1: Moderate Renal Impairment (Panel C): Participants with eGFR ≥30 - <60 mL/min/1.73 m² were enrolled in the Moderate Renal Impairment group.
- Part 1: Control to Match Panel C (Panel D): Participants with eGFR >/= 80 mL/min/1.73 m² were matched by age, gender, race, and body mass index (BMI) to participants in Panel C.
- Part 1: Severe Renal Impairment (Panel E): Participants with eGFR <30 mL/min/1.73 m² but not on dialysis were enrolled in the Severe Renal Impairment group.
- Part 1: Control to Match Panel E (Panel F): Participants with eGFR >/= 80 mL/min/1.73 m² were matched by age, gender, race, and body mass index (BMI) to participants in Panel E.
- Part 2: ESRD Requiring HD (Panel G): Participants with end-stage renal disease (ESRD) requiring hemodialysis (HD)
- Part 2: Control to Match Panel G (Panel H): Participants with eGFR >/= 80 mL/min/1.73 m² were matched by age, gender, race, and body mass index (BMI) to participants in Panel G.
Period: Overall Study
Arm/Group | Part 1: Mild Renal Impairment (Panel A) | Part 1: Control to Match Panel A (Panel B) | Part 1: Moderate Renal Impairment (Panel C) | Part 1: Control to Match Panel C (Panel D) | Part 1: Severe Renal Impairment (Panel E) | Part 1: Control to Match Panel E (Panel F) | Part 2: ESRD Requiring HD (Panel G) | Part 2: Control to Match Panel G (Panel H)
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Mild Renal Impairment (Panel A) | Part 1: Control to Match Panel A (Panel B) | Part 1: Moderate Renal Impairment (Panel C) | Part 1: Control to Match Panel C (Panel D) | Part 1: Severe Renal Impairment (Panel E) | Part 1: Control to Match Panel E (Panel F) | Part 2: ESRD Requiring HD (Panel G) | Part 2: Control to Match Panel G (Panel H) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 49
Age, Continuous [Mean (Full Range); unit: Years] | 71 [67 to 75] | 68 [64 to 74] | 62 [50 to 74] | 60 [51 to 74] | 64 [54 to 72] | 60 [51 to 69] | 46 [36 to 60] | 43 [33 to 57] | 59 [33 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 2 | 2 | 2 | 2 | 3 | 21
  Male | 2 | 2 | 4 | 4 | 4 | 4 | 4 | 4 | 28

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC0-∞) of Omarigliptin
Description: AUC0-∞ is a measure of the mean concentration levels of drug in the plasma after the dose.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 (Panel G only), 96, 168, 240, and 336 hours post-dose
Population: All participants that received a single 3 mg dose of omarigliptin.
Measure: Geometric Mean (95% Confidence Interval); unit: nM*hr
Groups:
- Part 2: ESRD Requiring HD (Panel G) - Period 1: Participants with end-stage renal disease (ESRD) requiring hemodialysis (HD) were enrolled in Panel G. In Period 1, participants received MK-3102 3 mg immediately after HD. One participant did not have an estimable parameter.
- Part 2: Control to Match Panel G (Panel H) - Period 1; Part 2: Control to Match Panel G (Panel H) - Period 2: Participants were matched by age, gender, race, and body mass index (BMI) to participants in Panel G. Data from the participant that withdrew from study was not included.
- Part 2: ESRD Requiring HD (Panel G) - Period 2: Participants with ESRD requiring HD were enrolled in Panel G. In Period 2, participants received MK-3102 3 mg 2 hours prior to HD.
Arm/Group | Part 1: Mild Renal Impairment (Panel A) | Part 1: Control to Match Panel A (Panel B) | Part 1: Moderate Renal Impairment (Panel C) | Part 1: Control to Match Panel C (Panel D) | Part 1: Severe Renal Impairment (Panel E) | Part 1: Control to Match Panel E (Panel F) | Part 2: ESRD Requiring HD (Panel G) - Period 1 | Part 2: Control to Match Panel G (Panel H) - Period 1 | Part 2: ESRD Requiring HD (Panel G) - Period 2 | Part 2: Control to Match Panel G (Panel H) - Period 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6
nM*hr | 4703.16 [4078.19 to 5423.92] | 4983.58 [4321.34 to 5747.31] | 5785.21 [4950.03 to 6761.31] | 4312.17 [3689.64 to 5039.74] | 6466.65 [5577.34 to 7497.76] | 4142.94 [3573.19 to 4803.53] | 7257.17 [5595.73 to 9411.93] | 3842.62 [2964.77 to 4980.39] | 7585.94 [5852.93 to 9832.07] | 3842.62 [2964.77 to 4980.39]
Statistical Analysis 1: Comparison: Part 1: Mild Renal Impairment (Panel A) vs Part 1: Control to Match Panel A (Panel B); Test type: Superiority or Other; Geometric mean ratio (GMR); GMR of Panel A:Panel B; GMR = 0.94, 90% CI 2-sided [0.80 to 1.11]
Statistical Analysis 2: Comparison: Part 1: Moderate Renal Impairment (Panel C) vs Part 1: Control to Match Panel C (Panel D); Test type: Superiority or Other; GMR of Panel C:Panel D; GMR of Panel C:Panel D = 1.34, 90% CI 2-sided [1.12 to 1.61]
Statistical Analysis 3: Comparison: Part 1: Severe Renal Impairment (Panel E) vs Part 1: Control to Match Panel E (Panel F); Test type: Superiority or Other; GMR of Panel E:Panel F; GMR of Panel E:Panel F = 1.56, 90% CI 2-sided [1.32 to 1.85]
Statistical Analysis 4: Comparison: Part 2: ESRD Requiring HD (Panel G) - Period 1 vs Part 2: Control to Match Panel G (Panel H) - Period 1; Test type: Superiority or Other; GMR of Panel G:Panel H; GMR or Panel G:Panel H = 1.89, 90% CI 2-sided [1.40 to 2.55]
Statistical Analysis 5: Comparison: Part 2: ESRD Requiring HD (Panel G) - Period 2 vs Part 2: Control to Match Panel G (Panel H) - Period 2; Test type: Superiority or Other; GMR of Panel G:Panel H; GMR of Panel G:Panel H = 1.97, 90% CI 2-sided [1.46 to 2.66]

2. Primary Outcome: Maximum Concentration (Cmax) of Omarigliptin
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 (Panel G only), 96, 168, 240, and 336 hours post-dose
Population: All participants that received a single 3 mg dose of omarigliptin.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Groups:
- Part 2: ESRD Requiring HD (Panel G) - Period 1: Participants with end-stage renal disease (ESRD) requiring hemodialysis (HD) were enrolled in Panel G. In Period 1, participants received MK-3102 3 mg immediately after HD.
- Part 2: Control to Match Panel G (Panel H) - Period 1; Part 2: Control to Match Panel G (Panel H) - Period 2: Participants were matched by age, gender, race, and body mass index (BMI) to participants in Panel G. Data from one participant who withdrew from study and data from the replacement participant are both included.
Arm/Group | Part 1: Mild Renal Impairment (Panel A) | Part 1: Control to Match Panel A (Panel B) | Part 1: Moderate Renal Impairment (Panel C) | Part 1: Control to Match Panel C (Panel D) | Part 1: Severe Renal Impairment (Panel E) | Part 1: Control to Match Panel E (Panel F) | Part 2: ESRD Requiring HD (Panel G) - Period 1 | Part 2: Control to Match Panel G (Panel H) - Period 1 | Part 2: ESRD Requiring HD (Panel G) - Period 2 | Part 2: Control to Match Panel G (Panel H) - Period 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 6 | 7
nM | 60.37 (51.82) [51.82 to 70.34] | 64.03 [54.96 to 74.61] | 61.43 [50.64 to 74.52] | 54.34 [44.80 to 65.92] | 48.65 [37.29 to 63.48] | 53.89 [41.30 to 70.31] | 41.43 [32.67 to 52.54] | 56.06 [44.99 to 69.85] | 40.98 [32.31 to 51.97] | 56.06 [44.99 to 69.85]
Statistical Analysis 1: Comparison: Part 1: Mild Renal Impairment (Panel A) vs Part 1: Control to Match Panel A (Panel B); Test type: Superiority or Other; GMR of Panel A:Panel B; GMR of Panel A:Panel B = 0.94, 90% CI 2-sided [0.79 to 1.12]
Statistical Analysis 2: Comparison: Part 1: Moderate Renal Impairment (Panel C) vs Part 1: Control to Match Panel C (Panel D); Test type: Superiority or Other; GMR of Panel C:Panel D; GMR of Panel C:Panel D = 1.13, 90% CI 2-sided [0.91 to 1.41]
Statistical Analysis 3: Comparison: Part 1: Severe Renal Impairment (Panel E) vs Part 1: Control to Match Panel E (Panel F); Test type: Superiority or Other; GMR of Panel E:Panel F; GMR of Panel E:Panel F = 0.90, 90% CI 2-sided [0.66 to 1.23]
Statistical Analysis 4: Comparison: Part 2: ESRD Requiring HD (Panel G) - Period 1 vs Part 2: Control to Match Panel G (Panel H) - Period 1; Test type: Superiority or Other; GMR of Panel E:Panel F; GMR of Panel E:Panel F = 0.74, 90% CI 2-sided [0.57 to 0.96]
Statistical Analysis 5: Comparison: Part 2: ESRD Requiring HD (Panel G) - Period 2 vs Part 2: Control to Match Panel G (Panel H) - Period 2; Test type: Superiority or Other; GMR of Panel E:Panel F; GMR of Panel E:Panel F = 0.73, 90% CI 2-sided [0.56 to 0.95]

3. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to 168 Hours Post Dose (AUC0-168h) of Omarigliptin
Description: AUC0-168h is a measure of the total amount of drug in the plasma from the dose to 168 hours after the dose.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 (Panel G only), 96, and 168 hours post-dose
Population: All participants that received a single 3 mg dose of omarigliptin.
Measure: Geometric Mean (95% Confidence Interval); unit: nM*hr
Arm/Group | Part 1: Mild Renal Impairment (Panel A) | Part 1: Control to Match Panel A (Panel B) | Part 1: Moderate Renal Impairment (Panel C) | Part 1: Control to Match Panel C (Panel D) | Part 1: Severe Renal Impairment (Panel E) | Part 1: Control to Match Panel E (Panel F) | Part 2: ESRD Requiring HD (Panel G) - Period 1 | Part 2: Control to Match Panel G (Panel H) - Period 1 | Part 2: ESRD Requiring HD (Panel G) - Period 2 | Part 2: Control to Match Panel G (Panel H) - Period 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 6 | 7
nM*hr | 3055.48 [2720.74 to 3431.42] | 3315.01 [2951.83 to 3722.87] | 3674.50 [3037.78 to 4444.68] | 2770.54 [2290.46 to 3351.25] | 3580.02 [3040.51 to 4215.27] | 2615.56 [2221.40 to 3079.67] | 3352.27 [2653.44 to 4235.17] | 2431.77 [1958.50 to 3019.41] | 3150.93 [2494.07 to 3980.80] | 2431.77 [1958.50 to 3019.41]
Statistical Analysis 1: Comparison: Part 1: Mild Renal Impairment (Panel A) vs Part 1: Control to Match Panel A (Panel B); Test type: Superiority or Other; GMR of Panel A:Panel B; GMR of Panel A:Panel B = 0.92, 90% CI 2-sided [0.81 to 1.05]
Statistical Analysis 2: Comparison: Part 1: Moderate Renal Impairment (Panel C) vs Part 1: Control to Match Panel C (Panel D); Test type: Superiority or Other; GMR of Panel C:Panel D; GMR of Panel C:Panel D = 1.33, 90% CI [1.07 to 1.65]
Statistical Analysis 3: Comparison: Part 1: Severe Renal Impairment (Panel E) vs Part 1: Control to Match Panel E (Panel F); Test type: Superiority or Other; GMR of Panel E:Panel F; GMR of Panel E:Panel F = 1.37, 90% CI 2-sided [1.13 to 1.65]
Statistical Analysis 4: Comparison: Part 2: ESRD Requiring HD (Panel G) - Period 1 vs Part 2: Control to Match Panel G (Panel H) - Period 1; Test type: Superiority or Other; GMR of Panel G:Panel H; GMR of Panel G:Panel H = 1.38, 90% CI 2-sided [1.06 to 1.79]
Statistical Analysis 5: Comparison: Part 2: ESRD Requiring HD (Panel G) - Period 2 vs Part 2: Control to Match Panel G (Panel H) - Period 2; Test type: Superiority or Other; GMR of Panel G:Panel H; GMR of Panel G:Panel H = 1.30, 90% CI 2-sided [1.00 to 1.68]

4. Primary Outcome: Concentration at 168 Hours Post-dose (C168h) of Omarigliptin
Description: C168h is a measure of the plasma drug concentration 168 hours post-dose.
Time Frame: 168 hours post-dose
Population: All participants that received a single 3 mg dose of omarigliptin.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Part 1: Mild Renal Impairment (Panel A) | Part 1: Control to Match Panel A (Panel B) | Part 1: Moderate Renal Impairment (Panel C) | Part 1: Control to Match Panel C (Panel D) | Part 1: Severe Renal Impairment (Panel E) | Part 1: Control to Match Panel E (Panel F) | Part 2: ESRD Requiring HD (Panel G) - Period 1 | Part 2: Control to Match Panel G (Panel H) - Period 1 | Part 2: ESRD Requiring HD (Panel G) - Period 2 | Part 2: Control to Match Panel G (Panel H) - Period 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 6 | 7
nM | 7.19 [6.06 to 8.53] | 7.85 [6.62 to 9.31] | 9.10 [7.68 to 10.78] | 6.28 [5.30 to 7.44] | 11.48 [9.64 to 13.69] | 6.28 [5.27 to 7.49] | 11.46 [8.81 to 14.91] | 6.05 [4.74 to 7.71] | 11.35 [8.72 to 14.76] | 6.05 [4.74 to 7.71]
Statistical Analysis 1: Comparison: Part 1: Mild Renal Impairment (Panel A) vs Part 1: Control to Match Panel A (Panel B); Test type: Superiority or Other; GMR of Panel A:Panel B; GMR of Panel A:Panel B = 0.92, 90% CI 2-sided [0.75 to 1.12]
Statistical Analysis 2: Comparison: Part 1: Moderate Renal Impairment (Panel C) vs Part 1: Control to Match Panel C (Panel D); Test type: Superiority or Other; GMR of Panel C:Panel D; GMR of Panel C:Panel D = 1.45, 90% CI 2-sided [1.19 to 1.76]
Statistical Analysis 3: Comparison: Part 1: Severe Renal Impairment (Panel E) vs Part 1: Control to Match Panel E (Panel F); Test type: Superiority or Other; GMR of Panel E:Panel F; GMR of Panel E:Panel F = 1.83, 90% CI 2-sided [1.49 to 2.24]
Statistical Analysis 4: Comparison: Part 2: ESRD Requiring HD (Panel G) - Period 1 vs Part 2: Control to Match Panel G (Panel H) - Period 1; Test type: Superiority or Other; GMR of Panel G:Panel H; GMR of Panel G:Panel H = 1.90, 90% CI 2-sided [1.41 to 2.54]
Statistical Analysis 5: Comparison: Part 2: ESRD Requiring HD (Panel G) - Period 2 vs Part 2: Control to Match Panel G (Panel H) - Period 2; Test type: Superiority or Other; GMR of Panel G:Panel H; GMR of Panel G:Panel H = 1.88, 90% CI 2-sided [1.40 to 2.52]

5. Primary Outcome: Apparent Volume of Distribution (Vd/F) of Omarigliptin
Description: Vd/F is defined as the distribution of a medication between the plasma and the rest of the body after the dose. It is the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of the drug.
Time Frame: Up to 336 hours post-dose
Population: All participants that received a single 3 mg dose of omarigliptin.
Measure: Geometric Mean (95% Confidence Interval); unit: L
Groups:
- Part 2: Control to Match Panel G (Panel H) - Period 2: Participants were matched by age, gender, race, and body mass index (BMI) to participants in Panel G. Data from the participant that withdrew from the study was not included.
Arm/Group | Part 1: Mild Renal Impairment (Panel A) | Part 1: Control to Match Panel A (Panel B) | Part 1: Moderate Renal Impairment (Panel C) | Part 1: Control to Match Panel C (Panel D) | Part 1: Severe Renal Impairment (Panel E) | Part 1: Control to Match Panel E (Panel F) | Part 2: ESRD Requiring HD (Panel G) - Period 1 | Part 2: Control to Match Panel G (Panel H) - Period 1 | Part 2: ESRD Requiring HD (Panel G) - Period 2 | Part 2: Control to Match Panel G (Panel H) - Period 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6
L | 349.42 [282.17 to 432.69] | 314.39 [253.88 to 389.31] | 295.86 [218.39 to 400.82] | 392.75 [289.90 to 532.08] | 280.58 [216.30 to 363.95] | 410.21 [316.24 to 532.11] | 334.57 [249.27 to 449.07] | 478.52 [357.04 to 641.32] | 383.12 [285.87 to 513.47] | 478.52 [357.04 to 641.32]
Statistical Analysis 1: Comparison: Part 1: Mild Renal Impairment (Panel A) vs Part 1: Control to Match Panel A (Panel B); Test type: Superiority or Other; GMR of Panel A:Panel B; GMR of Panel A:Panel B = 1.11, 90% CI 2-sided [0.87 to 1.42]
Statistical Analysis 2: Comparison: Part 1: Moderate Renal Impairment (Panel C) vs Part 1: Control to Match Panel C (Panel D); Test type: Superiority or Other; GMR of Panel C:Panel D; GMR of Panel C:Panel D = 0.75, 90% CI 2-sided [0.53 to 1.07]
Statistical Analysis 3: Comparison: Part 1: Severe Renal Impairment (Panel E) vs Part 1: Control to Match Panel E (Panel F); Test type: Superiority or Other; GMR of Panel E:Panel F; GMR of Panel E:Panel F = 0.68, 90% CI 2-sided [0.51 to 0.92]
Statistical Analysis 4: Comparison: Part 2: ESRD Requiring HD (Panel G) - Period 1 vs Part 2: Control to Match Panel G (Panel H) - Period 1; Test type: Superiority or Other; GMR of Panel G:Panel H; GMR of Panel G:Panel H = 0.70, 90% CI 2-sided [0.50 to 0.98]
Statistical Analysis 5: Comparison: Part 2: ESRD Requiring HD (Panel G) - Period 2 vs Part 2: Control to Match Panel G (Panel H) - Period 2; Test type: Superiority or Other; GMR of Panel G:Panel H; GMR of Panel G:Panel H = 0.80, 90% CI 2-sided [0.57 to 1.12]

6. Primary Outcome: Apparent Total Body Clearance (CL/F) of Omarigliptin
Description: CL/F is a calculation of the rate at which a drug is removed from the body via renal, hepatic, and other clearance pathways, expressed as volume (milliliters) per unit of time (minutes).
Time Frame: Up to 336 hours post-dose
Population: All participants that received a single 3 mg dose of omarigliptin.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Part 1: Mild Renal Impairment (Panel A) | Part 1: Control to Match Panel A (Panel B) | Part 1: Moderate Renal Impairment (Panel C) | Part 1: Control to Match Panel C (Panel D) | Part 1: Severe Renal Impairment (Panel E) | Part 1: Control to Match Panel E (Panel F) | Part 2: ESRD Requiring HD (Panel G) - Period 1 | Part 2: Control to Match Panel G (Panel H) - Period 1 | Part 2: ESRD Requiring HD (Panel G) - Period 2 | Part 2: Control to Match Panel G (Panel H) - Period 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6
mL/min | 26.51 [22.98 to 30.57] | 25.02 [21.69 to 28.85] | 21.55 [18.44 to 25.18] | 28.91 [24.74 to 33.79] | 19.28 [16.63 to 22.35] | 30.09 [25.95 to 34.89] | 17.18 [13.25 to 22.28] | 32.44 [25.03 to 42.05] | 16.43 [12.68 to 21.30] | 32.44 [25.03 to 42.05]
Statistical Analysis 1: Comparison: Part 1: Mild Renal Impairment (Panel A) vs Part 1: Control to Match Panel A (Panel B); Test type: Superiority or Other; GMR of Panel A:Panel B; GMR of Panel A:Panel B = 1.06, 90% CI 2-sided [0.90 to 1.25]
Statistical Analysis 2: Comparison: Part 1: Moderate Renal Impairment (Panel C) vs Part 1: Control to Match Panel C (Panel D); Test type: Superiority or Other; GMR of Panel C:Panel D; GMR of Panel C:Panel D = 0.75, 90% CI 2-sided [0.62 to 0.89]
Statistical Analysis 3: Comparison: Part 1: Severe Renal Impairment (Panel E) vs Part 1: Control to Match Panel E (Panel F); Test type: Superiority or Other; GMR of Panel E:Panel F; GMR of Panel E:Panel F = 0.64, 90% CI 2-sided [0.54 to 0.76]
Statistical Analysis 4: Comparison: Part 2: ESRD Requiring HD (Panel G) - Period 1 vs Part 2: Control to Match Panel G (Panel H) - Period 1; Test type: Superiority or Other; GMR of Panel G:Panel H; GMR of Panel G:Panel H = 0.53, 90% CI 2-sided [0.39 to 0.71]
Statistical Analysis 5: Comparison: Part 2: ESRD Requiring HD (Panel G) - Period 2 vs Part 2: Control to Match Panel G (Panel H) - Period 2; Test type: Superiority or Other; GMR of Panel G:Panel H; GMR of Panel G:Panel H = 0.51, 90% CI 2-sided [0.38 to 0.68]

7. Primary Outcome: Renal Clearance (CLr) of Omarigliptin
Description: CLr is a calculation of the rate at which a drug is removed from the body via renal clearance pathways, expressed as volume (milliliters) per unit of time (minutes). CLr was only determined for Panels A-F.
Time Frame: Up to 336 hours post-dose
Population: All participants that received a single 3 mg dose of omarigliptin.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Part 1: Mild Renal Impairment (Panel A) | Part 1: Control to Match Panel A (Panel B) | Part 1: Moderate Renal Impairment (Panel C) | Part 1: Control to Match Panel C (Panel D) | Part 1: Severe Renal Impairment (Panel E) | Part 1: Control to Match Panel E (Panel F)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
mL/min | 27.26 [22.25 to 33.41] | 29.27 [23.89 to 35.87] | 17.93 [14.06 to 22.87] | 24.71 [19.37 to 31.52] | 12.18 [9.79 to 15.14] | 28.84 [23.19 to 35.86]
Statistical Analysis 1: Comparison: Part 1: Mild Renal Impairment (Panel A) vs Part 1: Control to Match Panel A (Panel B); Test type: Superiority or Other; GMR of Panel A:Panel B; GMR of Panel A:Panel B = 0.93, 90% CI 2-sided [0.74 to 1.18]
Statistical Analysis 2: Comparison: Part 1: Moderate Renal Impairment (Panel C) vs Part 1: Control to Match Panel C (Panel D); Test type: Superiority or Other; GMR of Panel C:Panel D; GMR of Panel C:Panel D = 0.73, 90% CI 2-sided [0.55 to 0.96]
Statistical Analysis 3: Comparison: Part 1: Severe Renal Impairment (Panel E) vs Part 1: Control to Match Panel E (Panel F); Test type: Superiority or Other; GMR of Panel E:Panel F; GMR of Panel E:Panel F = 0.42, 90% CI 2-sided [0.33 to 0.54]

8. Primary Outcome: Fraction of Dose Excreted Unchanged in Urine Through 48 Hours Post-dose (fe48h) of Omarigliptin
Description: fe48h is expressed as percentage of omarigliptin not metabolized and excreted in urine. fe48h was only determined for Panels A-F.
Time Frame: Up to 48 hours post-dose
Population: All participants that received a single 3 mg dose of omarigliptin.
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage of total dose
Arm/Group | Part 1: Mild Renal Impairment (Panel A) | Part 1: Control to Match Panel A (Panel B) | Part 1: Moderate Renal Impairment (Panel C) | Part 1: Control to Match Panel C (Panel D) | Part 1: Severe Renal Impairment (Panel E) | Part 1: Control to Match Panel E (Panel F)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Percentage of total dose | 35 [29 to 43] | 41 [34 to 50] | 27 [22 to 33] | 30 [24 to 37] | 15 [12 to 20] | 31 [24 to 40]
Statistical Analysis 1: Comparison: Part 1: Mild Renal Impairment (Panel A) vs Part 1: Control to Match Panel A (Panel B); Test type: Superiority or Other; GMR of Panel A:Panel B; GMR of Panel A:Panel B = 0.86, 90% CI 2-sided [0.69 to 1.07]
Statistical Analysis 2: Comparison: Part 1: Moderate Renal Impairment (Panel C) vs Part 1: Control to Match Panel C (Panel D); Test type: Superiority or Other; GMR of Panel C:Panel D; GMR of Panel C:Panel D = 0.90, 90% CI 2-sided [0.70 to 1.15]
Statistical Analysis 3: Comparison: Part 1: Severe Renal Impairment (Panel E) vs Part 1: Control to Match Panel E (Panel F); Test type: Superiority or Other; GMR of Panel E:Panel F; GMR of Panel E:Panel F = 0.50, 90% CI 2-sided [0.37 to 0.67]

9. Primary Outcome: Cumulative Amount of Drug Excreted in Urine Over 48 Hours (Ae0-48h) of Omarigliptin
Description: Ae0-48h is a measure of the cumulative amount of drug excreted in the urine for 48 hours post-dose. Ae0-48h was only determined for Panels A-F.
Time Frame: Up to 48 hours post-dose
Population: All participants that received a single 3 mg dose of omarigliptin.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg
Arm/Group | Part 1: Mild Renal Impairment (Panel A) | Part 1: Control to Match Panel A (Panel B) | Part 1: Moderate Renal Impairment (Panel C) | Part 1: Control to Match Panel C (Panel D) | Part 1: Severe Renal Impairment (Panel E) | Part 1: Control to Match Panel E (Panel F)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
mg | 1.04 [0.86 to 1.25] | 1.21 [1.00 to 1.46] | 0.79 [0.64 to 0.98] | 0.88 [0.71 to 1.10] | 0.45 [0.35 to 0.58] | 0.90 [0.70 to 1.16]
Statistical Analysis 1: Comparison: Part 1: Mild Renal Impairment (Panel A) vs Part 1: Control to Match Panel A (Panel B); Test type: Superiority or Other; GMR of Panel A:Panel B; GMR of Panel A:Panel B = 0.86, 90% CI 2-sided [0.69 to 1.07]
Statistical Analysis 2: Comparison: Part 1: Moderate Renal Impairment (Panel C) vs Part 1: Control to Match Panel C (Panel D); Test type: Superiority or Other; GMR of Panel C:Panel D; GMR of Panel C:Panel D = 0.90, 90% CI 2-sided [0.70 to 1.15]
Statistical Analysis 3: Comparison: Part 1: Severe Renal Impairment (Panel E) vs Part 1: Control to Match Panel E (Panel F); Test type: Superiority or Other; GMR of Panel E:Panel F; GMR of Panel E:Panel F = 0.50, 90% CI 2-sided [0.37 to 0.67]

10. Primary Outcome: Time to Maximum Concentration (Tmax) of Omarigliptin
Description: Tmax is a measure of the time to reach the maximum drug plasma concentration post-dose.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 (Panel G only), 96, 168, 240, and 336 hours post-dose
Population: All participants that received a single 3 mg dose of omarigliptin.
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: Mild Renal Impairment (Panel A) | Part 1: Control to Match Panel A (Panel B) | Part 1: Moderate Renal Impairment (Panel C) | Part 1: Control to Match Panel C (Panel D) | Part 1: Severe Renal Impairment (Panel E) | Part 1: Control to Match Panel E (Panel F) | Part 2: ESRD Requiring HD (Panel G) - Period 1 | Part 2: Control to Match Panel G (Panel H) - Period 1 | Part 2: ESRD Requiring HD (Panel G) - Period 2 | Part 2: Control to Match Panel G (Panel H) - Period 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 6 | 7
hour | 3.0 [1.0 to 4.0] | 1.5 [1.0 to 4.0] | 2.0 [1.0 to 6.0] | 1.5 [1.0 to 2.0] | 2.0 [1.0 to 6.0] | 1.5 [1.0 to 2.0] | 4.0 [2.0 to 6.0] | 1.0 [0.5 to 4.0] | 4.0 [1.0 to 6.2] | 1.0 [0.5 to 4.0]

11. Primary Outcome: Apparent Terminal Half-life (t1/2) of Omarigliptin
Description: T1/2 is the time required for the maximum concentration of a drug in the plasma to decrease by 50%.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 (Panel G only), 96, 168, 240, and 336 hours post-dose
Population: All participants that received a single 3 mg dose of omarigliptin.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part 1: Mild Renal Impairment (Panel A) | Part 1: Control to Match Panel A (Panel B) | Part 1: Moderate Renal Impairment (Panel C) | Part 1: Control to Match Panel C (Panel D) | Part 1: Severe Renal Impairment (Panel E) | Part 1: Control to Match Panel E (Panel F) | Part 2: ESRD Requiring HD (Panel G) - Period 1 | Part 2: Control to Match Panel G (Panel H) - Period 1 | Part 2: ESRD Requiring HD (Panel G) - Period 2 | Part 2: Control to Match Panel G (Panel H) - Period 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6
hour | 148.3 (39.0) | 143.7 (21.9) | 156.2 (32.0) | 147.0 (65.4) | 159.8 (55.7) | 155.0 (33.5) | 215.4 (38.7) | 162.6 (53.7) | 263.7 (62.7) | 162.6 (53.7)

12. Secondary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure (signs), function (symptoms), or chemistry (laboratory data) of the body temporally associated with any use of a Sponsor product, whether or not considered related to the use of the product.
Time Frame: From pre-dose to 14 days post-dose (Up to Day 15)
Population: All participants that received a single 3 mg dose of omarigliptin.
Measure: Number; unit: Participants
Groups:
- Part 2: ESRD Requiring HD (Panel G) - Periods 1 and 2: Participants with end-stage renal disease (ESRD) requiring hemodialysis (HD) were enrolled in Panel G.
Arm/Group | Part 1: Mild Renal Impairment (Panel A) | Part 1: Control to Match Panel A (Panel B) | Part 1: Moderate Renal Impairment (Panel C) | Part 1: Control to Match Panel C (Panel D) | Part 1: Severe Renal Impairment (Panel E) | Part 1: Control to Match Panel E (Panel F) | Part 2: ESRD Requiring HD (Panel G) - Periods 1 and 2 | Part 2: Control to Match Panel G (Panel H) - Period 1
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7
Participants | 1 | 1 | 4 | 1 | 1 | 1 | 0 | 1

13. Secondary Outcome: Number of Participants Withdrawn From Study
Time Frame: Up to Day 15
Population: All participants that received a single 3 mg dose of omarigliptin.
Measure: Number; unit: Participants
Arm/Group | Part 1: Mild Renal Impairment (Panel A) | Part 1: Control to Match Panel A (Panel B) | Part 1: Moderate Renal Impairment (Panel C) | Part 1: Control to Match Panel C (Panel D) | Part 1: Severe Renal Impairment (Panel E) | Part 1: Control to Match Panel E (Panel F) | Part 2: ESRD Requiring HD (Panel G) - Periods 1 and 2 | Part 2: Control to Match Panel G (Panel H) - Period 1
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From pre-dose to 14 days post-dose (up to Day 15)
Description: An adverse experience is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the Sponsor's product, whether or not considered related to the use of the product.
Groups:
- Part 2: Control to Match Panel G (Panel H): Participants with eGFR >/= 80 mL/min/1.73 m² were matched by age, gender, race, and body mass index (BMI) to participants in Panel G. Data from one participant who withdrew from study and data from the replacement participant are both included.
Arm/Group | Part 1: Mild Renal Impairment (Panel A) | Part 1: Control to Match Panel A (Panel B) | Part 1: Moderate Renal Impairment (Panel C) | Part 1: Control to Match Panel C (Panel D) | Part 1: Severe Renal Impairment (Panel E) | Part 1: Control to Match Panel E (Panel F) | Part 2: ESRD Requiring HD (Panel G) | Part 2: Control to Match Panel G (Panel H)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 4/6 | 1/6 | 1/6 | 1/6 | 0/6 | 1/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Mild Renal Impairment (Panel A) (N=6) | Part 1: Control to Match Panel A (Panel B) (N=6) | Part 1: Moderate Renal Impairment (Panel C) (N=6) | Part 1: Control to Match Panel C (Panel D) (N=6) | Part 1: Severe Renal Impairment (Panel E) (N=6) | Part 1: Control to Match Panel E (Panel F) (N=6) | Part 2: ESRD Requiring HD (Panel G) (N=6) | Part 2: Control to Match Panel G (Panel H) (N=7)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eccymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.